CLINICAL TRIAL: NCT02382068
Title: Prevention of Cisplatin-Induced Ototoxicity by Intratympanic Dexamethasone
Brief Title: Dexamethasone in Preventing Hearing Loss in Patients Receiving Cisplatin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were enrolled to trial
Sponsor: Aaron Moberly (Other)
Responsible Party: Sponsor-Investigator, Aaron Moberly, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-12003; NCI-2014-01247 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-02-16; First posted 2015-03-06 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Malignant Neoplasm; Ototoxicity
MeSH Terms: conditions — Neoplasms; Ototoxicity | interventions — Dexamethasone; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (intratympanic dexamethasone) (Experimental): Patients receive dexamethasone via intratympanic injection in one ear and placebo via intratympanic injection in the other ear. Cisplatin standard of care treatment.
  Interventions: Drug: Dexamethasone; Other: Placebo; Drug: Cisplatin

INTERVENTIONS:
Drug: Dexamethasone — Given via intratympanic injection
  Other Names: DM
Other: Placebo — Given via intratympanic injection
  Other Names: PLCB
Drug: Cisplatin — Standard of care treatment with the following treatment course criteria:
  1. Dose: > 50 mg/m2
  2. Frequency: q3 -q4 weeks
  3. Cycles: 7 maximum
  Other Names: Platinol

SUMMARY:
This randomized pilot clinical trial studies dexamethasone in preventing hearing loss in patients receiving cisplatin. Injecting a steroid, such as dexamethasone, behind the eardrum before chemotherapy may help protect against cisplatin-associated hearing loss.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the potential protective effect of intratympanic dexamethasone administration on cisplatin-induced ototoxicity.

OUTLINE: Patients are randomized as to which ear receives dexamethasone.

Patients receive dexamethasone via intratympanic injection in one ear and placebo via intratympanic injection in the other ear.

After completion of study treatment, patients are followed up before each cisplatin treatment and then at 1 and 3 months after the last cisplatin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Planned cisplatin treatment restricted to the following treatment course criteria:

  * Dose: > 50 mg/m^2
  * Frequency: every (q)3-q4 weeks
  * Cycles: 7 maximum

Exclusion Criteria:

* Previous cisplatin treatment
* Previous or concurrent radiation treatment to the head and neck region
* Previous or existing pathology of the external or middle ear which would preclude auditory testing and/or intratympanic dexamethasone delivery
* Previous or existing pathology of the inner ear with or without hearing loss (i.e. sudden sensorineural hearing loss, Meniere's disease, autoimmune inner ear disease)
* Previous or existing pathology of the central nervous system with potential to impact auditory pathways (i.e. major head trauma, meningitis, encephalitis, brain metastasis, vestibular schwannoma)
* Recent steroid treatment within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in score of pure tone audiometry of conventional and high-frequency ranges (hearing level decibels [dB] hearing level) | Baseline to up to 3 months after completion of cisplatin treatment
  Change score will be assessed comparing baseline testing (prior to first cisplatin treatment) and various monitoring intervals (prior to each successive cisplatin treatment and 1 month and 3 months following completion of cisplatin treatment). Analyzed using a repeated measures model and a multi-level model.

SECONDARY OUTCOMES:
Change in score of distortion product otoacoustic emissions of conventional and high-frequency ranges (amplitude dB sound pressure level) | Baseline to up to 3 months after completion of cisplatin treatment
  Will be assessed comparing baseline testing (prior to first cisplatin treatment) and various monitoring intervals (prior to each successive cisplatin treatment and 1 months and 3 months following completion of cisplatin treatment). Analyzed using a repeated measures model and a multi-level model.
Presence of ototoxicity as defined by the American Speech-Language Hearing Association (ASHA) | Up to 3 months after completion of cisplatin treatment
  Presence or absence of ototoxicity as defined by the ASHA standards for pure tone audiometry (20 dB or greater change at any one test frequency, 10 dB or greater change at any two test frequencies, or any change at any three test frequencies). Analyzed using a repeated measures model and a multi-level model.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Moberly, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu